CLINICAL TRIAL: NCT01487603
Title: Feasibility of Evaluating Gene Alteration Analysis Using Samples Obtained by EBUS-TBNA in Patients With Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0109-CE
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
Keywords: Patients; undiagnosed enlarged; lymph nodes
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Tissue.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- confirmed or suspected lung cancer

SUMMARY:
Lung cancer is the leading cause of death in the world. Overall 5-year survival rate is fewer than 10% and the effectiveness of conventional chemotherapy is limited. The new knowledge shows the correlation between genetic alteration and effective of chemotherapy. Therefore non-surgical modalities to obtain tumor specimens for genetic alteration analysis are particularly critical in lung cancer, since many patients have advanced disease at the time of first presentation, and are therefore not eligible for radical surgery. Endobronchial ultrasound-guided transbronchial needle aspiration (EBUS-TBNA) samples obtained during diagnosis of lung cancer can be used for molecular analysis that will predict response to treatment and prognosis. In this study, we will detect specific target molecules related to the effectiveness of treatment (surgery, chemotherapy, radiotherapy) and prognosis in patients with lung cancer using EBUS-TBNA samples and its combined with xenograft technology.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Patients with confirmed or suspected lung cancer who require EBUS-TBNA as part of their staging investigations of the mediastinum will be considered for the trial.
* Patients with undiagnosed enlarged lymph nodes in the mediastinum suspicious for lung cancer in which a tissue diagnosis is required.

Exclusion Criteria:

* Patients who are deemed on clinical grounds not to be medically fit for a bronchoscopy.
* Patients where there is a high clinical suspicion of lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-10; Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to perform gene alteration analysis using samples obtained by EBUS-TBNA in lung cancer patients. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Yasufuku, MD, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada